CLINICAL TRIAL: NCT02074956
Title: A Phase I Randomized Placebo-Controlled, Double-Blind Study to Evaluate Safety and Immunogenicity of AERAS 404 When Administered as Different IC31 Adjuvant Amounts With Different AERAS-404 (HyVac4) Antigen Amounts in HIV-Negative BCG-Vaccinated Adults Without Evidence of Tuberculosis Infection
Brief Title: A Phase I Study to Evaluate Safety and Immunogenicity of AERAS 404 Administered in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C 006 404; C-006-404 (Other: Aeras)
Record Dates: First submitted 2014-02-27; First posted 2014-02-28 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Tuberculosis
Keywords: BCG Vaccinated; HIV Negative
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 AERAS-404 (Experimental): H4 Antigen at 5 ug IC31 Adjuvant 500 nmol
  2 doses at Study days 0 and 56
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 2 AERAS-404 (Experimental): H4 Antigen at 15 ug IC31 Adjuvant 500 nmol
  2 doses at Study days 0 and 56
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 3 AERAS-404 (Experimental): H4 Antigen at 50 ug IC31 Adjuvant 500 nmol
  2 doses at Study days 0 and 56
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 4 AERAS-404 (Experimental): H4 Antigen at 150 ug IC31 Adjuvant 500 nmol
  2 doses at Study days 0 and 56
  Interventions: Biological: AERAS-404; Biological: Placebo
- Cohort 5 AERAS-404 (Experimental): H4 Antigen at 5 ug or 15 ug IC31 Adjuvant 100 nmol Placebo - sterile buffer
  2 doses at Study days 0 and 56
  Interventions: Biological: AERAS-404; Biological: Placebo

INTERVENTIONS:
Biological: AERAS-404 — AERAS-404 is comprised of the H4 antigen, a fusion protein of Mycobacterium tuberculosis antigens 85B and TB10.4; and IC31 adjuvant, a combination of a leucine-rich peptide and a synthetic oligonucleotide.
  Other Names: H4
Biological: Placebo — Sterile buffer containing 10 mmol Tris and 169 mmol of NaCl in 0.8 mL of aqueous solution. This is the identical buffer solution in which H4 and IC31 are formulated.
  Other Names: Sterile Buffer

SUMMARY:
This Phase I study will be conducted as a randomized, double-blind, dose-escalation study in five groups of healthy adult male and female subjects who are BCG-vaccinated, HIV-negative, and have no evidence of tuberculosis infection. Since BCG-vaccinated individuals are the target population for which AERAS 404 might be indicated, AERAS 404 will be administered to individuals already vaccinated with BCG

DETAILED DESCRIPTION:
Sixty subjects will be sequentially enrolled into one of five study groups (i.e., Group 1, Group 2, Group 3, Group 4, or Group 5) with 10 subjects per group in Groups 1-4 and 20 subjects in Group 5. Within each study group, subjects will be randomized to a treatment assignment of either AERAS-404 or placebo control at a ratio of 4:1 (Groups 1-4) or two different dose amounts of AERAS-404 or placebo control at a ratio of 9:9:2 (Group 5) administered by intramuscular injection on Study Day 0 and Study Day 56. The principal investigator will determine an appropriate interval between the vaccinations such that the entire group is not dosed at the same time. All subjects will receive the same treatment on Study Day 0 as they receive on Study Day 56. All subjects will be followed for safety and immunogenicity evaluations for 182 days. A total of eleven clinic visits are planned (excluding screening) for all subjects

ELIGIBILITY:
Inclusion Criteria:

1. Has completed written informed consent
2. Is male or female
3. Is age 18 through 45 years on Study Day 0
4. Had BCG vaccination at least 5 years ago, documented through medical history or presence of scar
5. Has general good health, confirmed by medical history and physical examination
6. Has a Body Mass Index (BMI) between 19 and 33
7. Agrees to complete a follow-up period of 182 days as required by the protocol
8. Females: Agrees to avoid pregnancy from 28 days prior to Study Day 0 through the follow-up period of 182 days. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses) must agree to avoid pregnancy using an acceptable method
9. Agrees to avoid elective surgery for the duration of the study
10. Agrees to stay in contact with the investigative site for the study duration
11. Completed simultaneous enrollment in Aeras Vaccine Development Registry protocol

Exclusion Criteria:

1. Acute illness on Study Day 0
2. Axillary temperature >=37.5 degrees Celsius on Study Day 0
3. Evidence of significant active infection
4. Used immunosuppressive medication within 42 days before Study Day 0
5. Received immunoglobulin or blood products within 42 days before Study Day 0
6. Received any investigational drug therapy or investigational vaccine within 182 days before Study Day 0
7. Received inactivated influenza vaccine or inactivated tick-borne encephalitis vaccine within 14 days before entry into the study, or any other standard vaccine within 42 days before Study Day 0
8. Current chronic drug therapy including hormone replacement such as thyroxin, insulin
9. History or laboratory evidence of past, present or future possible immunodeficiency state which include any laboratory indication of HIV infection
10. History of allergic disease or reactions, including eczema
11. Previous medical history that may compromise safety of the subject in the study
12. Evidence of new acute illness that may compromise the safety of subject in the study
13. Evidence of chronic hepatitis
14. Inability to discontinue daily medications except contraceptives during study period
15. History of alcohol or drug abuse within past 2 years
16. Tobacco or cannabis smoking three or more days per week
17. Positive urine test for illicit drugs
18. History or evidence of any systemic disease on physical examination
19. History or evidence of active tuberculosis
20. Shared a residence within the last year with a individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis
21. All females: Positive urine pregnancy test during screening
22. Abnormal (per local laboratory parameters) chemistry and hematology parameters
23. QuantiFERON®-TB Gold evidence of Mtb infection
24. Received a tuberculin skin test within 3 months (90 days) prior to Study Day 0

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety profile of two injections of AERAS 404 at different dose levels of antigen and adjuvant. | Total duration of study follow up for all subjects is 182 days.
  Serious Adverse Events (SAE) will be collected on subjects throughout their participation in the study. Solicited and unsolicited adverse events are captured 28 days post each vaccination. The safety profile of AERAS-404 will be summarized by treatment regimen. The number (percentage) of subjects with adverse events will be summarized by MedDRA system organ class (SOC), and preferred term (PT). Additional summaries will present the number (percentage) of subjects with adverse events by severity and by relationship to study vaccine.

SECONDARY OUTCOMES:
Immunogenicity of two injections of AERAS 404 at different dose levels of antigen and adjuvant. | Immunogenicity was evaluated from blood collected at Study Days 0, 7, 14, 28, 56, 63, 70, 84, and 182. For all subjects, a QuantiFERON-TB Gold test was performed during screening and at Study Day 182
  Intracellular cytokine staining will be used to assess immunogenicity. Immune response based on percentages of CD4+ and CD8+ T cells that produced one, two, or three cytokines (IFN-γ, TNF-α, and/or IL-2) in response to stimulation with one of 2 antigenic peptide pools (Ag85B and TB10.4) derived from and representing the entire amino acid sequences of the mycobacterial antigens Ag85B and TB10.4, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongkai Shi, MD, Study Director — Aeras; Timo Vesikari, MD, Principal Investigator — University of Tampere Vaccine Research Clinic
Locations (1):
- University of Tampere Vaccine Research Clinic, Biokatu, Pirkanmaa, Finland

REFERENCES:
- [Derived] Norrby M, Vesikari T, Lindqvist L, Maeurer M, Ahmed R, Mahdavifar S, Bennett S, McClain JB, Shepherd BM, Li D, Hokey DA, Kromann I, Hoff ST, Andersen P, de Visser AW, Joosten SA, Ottenhoff THM, Andersson J, Brighenti S. Safety and immunogenicity of the novel H4:IC31 tuberculosis vaccine candidate in BCG-vaccinated adults: Two phase I dose escalation trials. Vaccine. 2017 Mar 14;35(12):1652-1661. doi: 10.1016/j.vaccine.2017.01.055. Epub 2017 Feb 17. PMID 28216183